CLINICAL TRIAL: NCT01076231
Title: Feasibility and PhaseI/II Trial of Preoperative Proton Beam Radiotherapy With Concurrent Chemotherapy for Resectable Stage IIIA or Superior Sulcus NSCLC
Brief Title: Proton Beam Radiation Therapy and Chemotherapy in Treating Patients With Stage III Non-Small Cell Lung Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 25508; NCI-2010-00251
Record Dates: First submitted 2010-02-23; First posted 2010-02-26 (Estimated); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-04

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Proton Therapy; Cisplatin; Etoposide; Podophyllotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo proton beam radiotherapy over 5.5-7.5 weeks. Patients receive concurrent chemotherapy comprising cisplatin IV on days 1, 8, 29, and 36 and etoposide IV on days 1-5 and days 29-33.Treatment continues in the absence of disease progression or unacceptable toxicity.
  Beginning 4-6 weeks after completion of chemoradiotherapy, patients may undergo surgical resection or additional chemoradiotherapy.
  Interventions: Radiation: proton beam radiation therapy; Drug: cisplatin; Drug: etoposide; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Radiation: proton beam radiation therapy
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP; Neoplatin; PDD
Drug: etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; epipodophyllotoxin; VePesid; VP-16; VP-16-213
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Specialized radiation therapy, such as proton beam radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue in patients with non-small cell lung cancer. Drugs used in chemotherapy, such as cisplatin and etoposide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving proton beam radiation therapy together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of proton beam radiation therapy when given together with cisplatin and etoposide and to see how well it works in treating patients with stage III non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess feasibility. (Phase I) II. To determine dose-limiting toxicity and maximum tolerated dose. (Phase I) III. To determine the pathologic CR rate. (Phase II)

SECONDARY OBJECTIVES:

I. To assess late complications from irradiation using proton beam therapy in place of conventional photon beam therapy. (Phase II) II. To assess acute side effects from irradiation using proton beam therapy in place of conventional photon beam therapy. (Phase II) III. To compare the dose distribution to tumor and surrounding normal structures using DVH's (Dose Volume Histograms) generated from the proton plan used to treat the patient and the photon plan generated for comparison purposes. (Phase II) IV. To determine progression-free survival (Phase II) and late toxicity.

OUTLINE: This is a phase I, dose-escalation study of proton beam radiation therapy followed by a phase II study.

Patients undergo proton beam radiotherapy over 5.5-7.5 weeks. Patients receive concurrent chemotherapy comprising cisplatin IV on days 1, 8, 29, and 36 and etoposide IV on days 1-5 and days 29-33.Treatment continues in the absence of disease progression or unacceptable toxicity.

Beginning 4-6 weeks after completion of chemoradiotherapy, patients may undergo surgical resection or additional chemoradiotherapy.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion

* Histologically confirmed diagnosis of NSCLC
* Stage IIIA or Potentially resectable superior sulcus tumors
* No evidence of distant metastatic disease as documented by MRI of the brain and PET/CT
* Patients must have a Karnofsky Performance Status of >= 60
* Patients must be able to provide informed consent
* WBC >= 4000/mm^3
* Platelets >= 100,000 mm^3
* Creatinine =< 1.2 mg/dl (urinary diversion is permitted to improve renal function)
* Patients must have bilirubin =< 1.5 mg/dl
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.); hysterectomy or menopause must be clinically documented
* Negative pregnancy test for women of child-bearing age

Exclusion

* Prior or simultaneous malignancies within the past two years (other than cutaneous squamous or basal cell carcinoma, melanoma in situ or thyroid carcinoma) [For pts that will be on definitive treatment study, otherwise delete for umbrella recurrent protocol]
* Pregnant women, women planning to become pregnant and women that are nursing
* Actively being treated on any other research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2016-12 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Shabason, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Simone CB 2nd, Yegya-Raman N, Manjunath S, Verma V, Shabason JE, Xu L, Cengel KA, Levin WP, Berman AT, Christodouleas JP, Aggarwal C, Cohen RB, Langer CJ, Pechet TT, Singhal S, Kucharczuk JC, Rengan R, Feigenberg SJ. Prospective Feasibility and Phase 1/2 Trial of Preoperative Proton Beam Therapy With Concurrent Chemotherapy for Resectable Stage IIIA or Superior Sulcus Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2023 Nov 1;117(3):683-689. doi: 10.1016/j.ijrobp.2023.05.016. Epub 2023 May 17. No abstract available. PMID 37201756

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Patients undergo proton beam radiotherapy over 5.5-7.5 weeks. Patients receive concurrent chemotherapy comprising cisplatin IV on days 1, 8, 29, and 36 and etoposide IV on days 1-5 and days 29-33.Treatment continues in the absence of disease progression or unacceptable toxicity.
  Beginning 4-6 weeks after completion of chemoradiotherapy, patients may undergo surgical resection or additional chemoradiotherapy.
  proton beam radiation therapy
  cisplatin: Given IV
  etoposide: Given IV
  therapeutic conventional surgery
Period: Overall Study
Arm/Group | Arm I
Started | 34
Completed | 0
Not Completed | 34

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.88 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Deemed Feasible to Receive Intervention
Description: Feasibility will be based on multiple radiation planning and treatment parameters. Study will be deemed feasible if all patients are deemed feasible.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 21
Participants | 21

2. Primary Outcome: Dose-limiting Toxicity
Description: DLT is defined as post-operative mortality (within 30 days of surgery) or any grade 3 or higher pneumonitis or any other grade 4 or higher toxicity which occurs during chemoradiation or within 90 days following the end of treatment, whichever is longer.
Time Frame: 90 Days
Population: 19 patients underwent surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 19
Participants | 0

3. Primary Outcome: Late Toxicity
Description: Late toxicity is defined as any grade 3 or higher pneumonitis or any grade 4 or higher toxicity which occurs more than 90 days after surgery or completion of treatment.
Time Frame: 4.5 Years
Population: 19 patients underwent surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 19
Participants | 0

4. Secondary Outcome: Pathologic CR Rate
Description: Pathologic CR rate is defined as the fraction of patients who undergo surgery and have no evidence of disease based on surgical pathology.
Time Frame: 90 days
Population: 19 patients underwent surgery
Measure: Number; unit: complete response rate percentage
Arm/Group | Arm I
Number analyzed (Participants) | 19
complete response rate percentage | 21

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 21/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=34)
(Metabolism and nutrition disorders) | 5
Lymphocyte count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=34)
(Gastrointestinal disorders) | 12
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 4
Constipation (Gastrointestinal disorders) | 9
Dermatitis radiation (Injury, poisoning and procedural complications) | 7
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Esophageal pain (Gastrointestinal disorders) | 3
Esophagitis (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 10
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Headache (Nervous system disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 5
Insomnia (Psychiatric disorders) | 3
Lymphocyte count decreased (Investigations) | 6
Nausea (Gastrointestinal disorders) | 5
Platelet count decreased (Investigations) | 5
White blood cell decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes